CLINICAL TRIAL: NCT01370772
Title: Phase II Multicentric, Randomized Trial, Exploring Intensified Rituximab Prephase Monotherapy Before Standard Fludarabine-Cyclophosphamide-Rituximab Regimen in Previously Untreated Symptomatic B-cell Chronic Lymphocytic Leukemia
Brief Title: Intensified Rituimab Prephase Before FCR in Untreated B-CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL 2010 FMP
Record Dates: First submitted 2011-05-23; First posted 2011-06-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia CLL
Keywords: B CLL; Fist line treatment
MeSH Terms: interventions — Rituximab; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard R-FC arm (Active Comparator): Standard R-FC arm 6 cycles every 28 days
  * Cycle 1:
    * Rituximab : 375 mg/m² i.v on day 1
    * Fludarabine : 40 mg/m² per os, days 2-4, repeated every 28 days
    * Cyclophosphamide : 250 mg/m² per os, days 2-4, repeated every 28 days For patients with Leucocyte count > 25* G/L : rituximab in two equal doses at D1, D2
  * Cycle 2-6:
    * Rituximab: 500 mg/m² i.v on day 1, repeated every 28 days
    * Fludarabine : 40 mg/m² per os, days 2-4, repeated every 28 days
    * Cyclophosphamide : 250 mg/m² per os, days 2-4, repeated every 28 days
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- DenseR-FC arm (Experimental): DenseR-FC arm =1 prephase R Dense course +6 R-FC courses
  * Prephase:
    - Rituximab: 500 mg on day 0, 2000 mg on days 1, 8, and D15 For patients with Leucocyte count > 25* G/L : rituximab 250 mg D-1, D0 prephase
  * Cycle 1-6 (cycle 1 beginning at D22):
    * Rituximab: 500 mg/m2 i.v on day 1, repeated every 28 days
    * Fludarabine : 40 mg/m² per os, days 2-4, repeated every 28 days
    * Cyclophosphamide : 250 mg/m² per os, days 2-4, repeated every 28 days
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Rituximab — * Cycle 1 Rituximab : 375 mg/m² i.v on day 1
  * Cycle 2-6 Rituximab:500 mg/m² i.v on day 1, repeated every 28 days
  Other Names: R
  Arms: Standard R-FC arm
Drug: Rituximab — * Prephase: Rituximab:500 mg on day 0, 2000 mg on days 1, 8, and D15
  * Cycle 1-6 cycle 1 beginning at D22: Rituximab: 500 mg/m2 i.v on day 1, repeated every 28 days
  Other Names: R
  Arms: DenseR-FC arm
Drug: Cyclophosphamide — •FCR Cycle 1-6: Cyclophosphamide : 250 mg/m² per os, days 2-4, repeated every 28 days
  Other Names: C
Drug: Fludarabine — FCR Cycle 1-6: Fludarabine :40 mg/m² per os, days 2-4, repeated every 28 days
  Other Names: F

SUMMARY:
Phase II, multicenter, randomized trial, exploring intensified Rituximab prephase monotherapy before standard Fludarabine-Cyclophosphamide-Rituximab FC-R regimen in previously untreated symptomatic B-cell chronic lymphocytic leukemia CLL.

A Study from the Goelams GCFLLCMW intergroup

DETAILED DESCRIPTION:
Young fit medically B Cell untreated patients Comparison between FCR treatment = 6 FCR cycles and a the addition of a prephase with R Dense treatment before the 6 FCR cycles.

ELIGIBILITY:
Inclusion criteria:

* Patient information and written informed consent
* 18 years < Age < 66 ans
* confirmed B-CLL Matutes score 4 or 5
* Binet stage C or Binet stage A and B with active disease could be considered for inclusion. For stage A with active disease an agreement of investigator coordinator is required.
* no prior treatment except steroids for less than 1 month (detail corticoid)
* No 17p deletion as assessed by FISH < 10 % positive nuclei
* Performance status ECOG < 2
* CIRS Cumulative Illness Rating Scale < 6

Exclusion criteria:

* Binet stage A without active disease according to IWCLL 2008 criteria
* Know HIV seropositivity
* Hepatitis B or C seropositivity unless clearly due to vaccination
* Life expectancy < 6 months
* Clinically significant auto-immune anemia
* Active second malignancy currently requiring treatment (except basal cell carcinoma in situ endometrial carcinoma and incidental prostate carcinoma) and/or less than 5 years CR after breast cancer
* Any severe co-morbid conditions such as Class III or IV heart failure, myocardial infarction within 6 months, unstable angina, ventricular tachyarythmias requiring ongoing treatment, severe chronic obstructive pulmonary disease with hypoxemia, uncontrolled diabetes mellitus, or uncontrolled hypertension
* Concomitant disease requiring prolonged use of corticosteroids > 1 month
* Known hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the study drugs According to the SmPC or investigator practice
* Contraindication to use of Rituximab
* Transformation to aggressive B-cell malignancy e.g. diffuse large cell lymphoma, Hodgkin lymphoma, or prolymphocytic leukaemia
* Active bacterial, viral or fungal infection
* Abnormal renal function with creatinine clearance < 60 ml/min calculated according to the Cockcroft and Gault formula
* Total bilirubin, gamma glutamyltransferase or transaminase levels > 2.5 ULN.
* Any coexisting medical or psychological condition that would preclude participation in the required study procedures
* Patient with mental deficiency preventing proper understanding of the requirements of treatment.
* Pregnant or breastfeeding women.
* Adult under law-control
* Fertile male and female patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study.
* No afiliate to social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
complete response rates according to IWCLL 2008 guidelines with undetectable minimal residual disease | 9 months
  CR MRD negative rate at 9 months = treatment evaluation surveillance of cumulative toxicities of high dose rituximab

SECONDARY OUTCOMES:
To determine and compare the progression free survival PFS | 3 years
evaluate the immunophenotypic response rate after high dose Rituximab alone prephase in DenseR-FC | 9 months
  Treatment evaluation
To evaluate FcyRs polymorphisms influence on clinical response | 9 months
  R Dense arm treatment evaluation
To determine the pharmacokinetics of rituximab and determine the PK-PD relationship of rituximab based on biomarkers. | 12 months
To evaluate the safety profile of higher doses of rituximab | 41
  5 months treatment and 36 months follow up
To determine the event-free survival EFS | 3 years
To determine and compare the disease-free survival DFS | 3 years
To determine the overall survival OS | 3 years
To determine the time to next treatment TTNT | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CARTRON, MD PD, Principal Investigator — French Innovative Leukemia Organisation; Stephane LEPRETRE, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (2):
- France (2):
  - Stephane LEPRETRE, Rouen, CLCC Henri Becquerel
  - Guillaume CARTRON, Montpellier, Regional University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duroux-Richard I, Gagez AL, Alaterre E, Letestu R, Khalifa O, Jorgensen C, Lepretre S, Tchernonog E, Moreaux J, Cartron G, Apparailly F. miRNA profile at diagnosis predicts treatment outcome in patients with B-chronic lymphocytic leukemia: A FILO study. Front Immunol. 2022 Oct 17;13:983771. doi: 10.3389/fimmu.2022.983771. eCollection 2022. PMID 36325355
- [Derived] Gagez AL, Duroux-Richard I, Lepretre S, Orsini-Piocelle F, Letestu R, De Guibert S, Tuaillon E, Leblond V, Khalifa O, Gouilleux-Gruart V, Banos A, Tournilhac O, Dupuis J, Jorgensen C, Cartron G, Apparailly F. miR-125b and miR-532-3p predict the efficiency of rituximab-mediated lymphodepletion in chronic lymphocytic leukemia patients. A French Innovative Leukemia Organization study. Haematologica. 2017 Apr;102(4):746-754. doi: 10.3324/haematol.2016.153189. Epub 2017 Jan 25. PMID 28126961
- [Derived] Tout M, Gagez AL, Lepretre S, Gouilleux-Gruart V, Azzopardi N, Delmer A, Mercier M, Ysebaert L, Laribi K, Gonzalez H, Paintaud G, Cartron G, Ternant D. Influence of FCGR3A-158V/F Genotype and Baseline CD20 Antigen Count on Target-Mediated Elimination of Rituximab in Patients with Chronic Lymphocytic Leukemia: A Study of FILO Group. Clin Pharmacokinet. 2017 Jun;56(6):635-647. doi: 10.1007/s40262-016-0470-8. PMID 27783363
- See also: FILO Website — http://www.filo-leucemie.org